CLINICAL TRIAL: NCT04557527
Title: Suprachoroidal Visco-buckling for the Treatment of Rhegmatogenous Retinal Detachment: A Randomized, Controlled, Feasibility Trial
Brief Title: Suprachoroidal Visco-buckling for the Treatment of Rhegmatogenous Retinal Detachment
Acronym: VIKING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Norfolk and Norwich University Trust Foundation (Unknown); St Thomas' Hospital, London (Other); University of Sunderland (Other); Moorfields Eye Hospital NHS Foundation Trust (Other); Mid and South Essex NHS Foundation Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 283518
Record Dates: First submitted 2020-09-09; First posted 2020-09-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Retinal Detachment With Break
Keywords: retinal detachment; vitrectomy; gas tamponnade; suprachoroidal buckle; viscobuckle; postoperative recovery
MeSH Terms: conditions — Retinal Detachment | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Patient will be recruited into
Masking Description: randomisation software
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Other): Pars plana vitrectomy, retinopexy with laser or cryotherapy, and intravitreal gas tamponade.
  Interventions: Procedure: Pars plana vitrectomy, laser or cryo retinopexy and intraocular gas tamponade
- treatment (Active Comparator): Pars plana vitrectomy, laser retinopexy, suprachoroidal viscobuckle.
  Interventions: Device: Suprachoroidal viscobuckle with 2.3% Sodium hyaluronate (Healon 5 Ophthalmic viscoelastic device)

INTERVENTIONS:
Procedure: Pars plana vitrectomy, laser or cryo retinopexy and intraocular gas tamponade — Conventional pars plana vitrectomy procedure is used to treat rhegmatogenous retinal detachment- laser or cryo retinopexy intraocular gas tamponade (SF6, C2F6 or C3F8) are chosen according to the number and size of the causative retinal break(s) and surgeons clinical judgement
  Arms: control
Device: Suprachoroidal viscobuckle with 2.3% Sodium hyaluronate (Healon 5 Ophthalmic viscoelastic device) — After drainage of subretinal fluid, approximately 0.5 ml of Healon 5 is injected in to the suprachoroidal space underlying the retinal break. Laser retinopexy is applied around the break .
  Arms: treatment

SUMMARY:
The study compares standard surgery for retinal detachment (RD) (vitrectomy, cryotherapy and gas) with a surgical variation that replaces the intraocular gas tamponade with suprachoroidal injection of viscoelastic underneath the break that caused the retinal detachment.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks, the eligible patients who have given written consent to the treatment will be randomized into treatment (vitrectomy, cryo and gas) or control (viscobuckle vitrectomy) group.

ELIGIBILITY:
Inclusion Criteria:

Patients requiring pars plana vitrectomy for the treatment of primary rhegmatogenous retinal detachment (RD) caused by a single break, or multiple breaks within one clock hour. The final determination of qualifying breaks is made at the time of surgery following 360-degree, internal, indented search using a wide-angle viewing system.

Exclusion Criteria:

* Hypersensitivity to hyaluronate or. HEALON5® PRO OVD
* Participation in another interventional study within 8 weeks of enrolment or planned to occur during this study.
* Bleeding disorders or the use of anticoagulants (such as warfarin, rivaroxaban) or dual anti-platelet drugs such as aspirin with clopidogrel. Monotherapy with low dose (≤100 mg) aspirin is permitted, and if clinically appropriate this should be stopped prior to surgery and recommenced only after satisfactory day 1 post-operative review.
* Unwilling, unable, or unlikely to return for scheduled follow-up for the duration of the trial.
* Any other condition that, in the opinion of the investigator, would prevent the participant from granting informed consent or complying with the protocol, such as dementia, mental illness, or serious systemic medical disease.

Study eye:

* Presence of proliferative vitreoretinopathy (PVR) or any tractional RD
* Previous vitreoretinal surgery, open-globe injury or endophthalmitis
* Aphakia
* Previous or current congenital cataract
* Previous or current suprachoroidal haemorrhage
* Congenital or acquired ocular, orbital or periocular abnormality that, in the opinion of the attending vitreoretinal surgeon, would preclude the safe delivery of Healon 5 into the suprachoroidal space (detail the specific reason for exclusion in the source documents)
* Presence of other ocular co-morbidity that, in the opinion of the investigator, is likely to prevent an accurate assessment of retinal attachment
* Current intraocular inflammation other than mild cellular activity thought to be secondary to RD
* Current ocular or periocular infection other than blepharitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
To establish if it is feasible to recruit, retain, and evaluate patients with RD into a larger randomised controlled trial of vitrectomy and suprachoroidal viscobuckle. | 2 years
  feasibility trial
To make a preliminary assessment of safety and efficacy of suprachoroidal viscobuckle. | 2 years
  feasibility trial

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Guy's & St. Thomas' Hospital NHS Foundatrion Trust, London, London
  - Sunderland Eye Infimary, Sunderland, Tyne and Wear
  - Moorfields Eye Hospital, London
  - King's College Hospital NHS Foundation Trust, London
  - Norfolk and Norwich University Foundation Trust, Norwich
  - Southend University Hospital NHS Foundation Trust, Southend

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boden KT, Januschowski K, Szurman P. [Suprachoroidal Hydrogel Buckle - a New Minimal-Invasive Technique in Treatment of Rhegmatogenous Retinal Detachment]. Klin Monbl Augenheilkd. 2019 Mar;236(3):308-312. doi: 10.1055/s-0043-102947. Epub 2017 Apr 4. German. PMID 28376555
- [Background] El Rayes EN, Mikhail M, El Cheweiky H, Elsawah K, Maia A. SUPRACHOROIDAL BUCKLING FOR THE MANAGEMENT OF RHEGMATOGENOUS RETINAL DETACHMENTS SECONDARY TO PERIPHERAL RETINAL BREAKS. Retina. 2017 Apr;37(4):622-629. doi: 10.1097/IAE.0000000000001214. PMID 27482642
- [Background] Mikhail M, El-Rayes EN, Kojima K, Ajlan R, Rezende F. Catheter-guided suprachoroidal buckling of rhegmatogenous retinal detachments secondary to peripheral retinal breaks. Graefes Arch Clin Exp Ophthalmol. 2017 Jan;255(1):17-23. doi: 10.1007/s00417-016-3530-8. Epub 2016 Nov 16. PMID 27853956
- [Background] Mitry D, Awan MA, Borooah S, Siddiqui MA, Brogan K, Fleck BW, Wright A, Campbell H, Singh J, Charteris DG, Yorston D. Surgical outcome and risk stratification for primary retinal detachment repair: results from the Scottish Retinal Detachment study. Br J Ophthalmol. 2012 May;96(5):730-4. doi: 10.1136/bjophthalmol-2011-300581. Epub 2012 Jan 18. PMID 22257789
- [Background] Jackson TL, Donachie PH, Sallam A, Sparrow JM, Johnston RL. United Kingdom National Ophthalmology Database study of vitreoretinal surgery: report 3, retinal detachment. Ophthalmology. 2014 Mar;121(3):643-8. doi: 10.1016/j.ophtha.2013.07.015. Epub 2013 Aug 23. PMID 23978624
- [Background] Poole TA, Sudarsky RD. Suprachoroidal implantation for the treatment of retinal detachment. Ophthalmology. 1986 Nov;93(11):1408-12. doi: 10.1016/s0161-6420(86)33553-x. PMID 3808600
- [Background] Mohamed YH, Ono K, Kinoshita H, Uematsu M, Tsuiki E, Fujikawa A, Kitaoka T. Success Rates of Vitrectomy in Treatment of Rhegmatogenous Retinal Detachment. J Ophthalmol. 2016;2016:2193518. doi: 10.1155/2016/2193518. Epub 2016 Jul 13. PMID 27478632